CLINICAL TRIAL: NCT03040843
Title: Documentation of Altered Mental Status
Status: Completed | Type: Observational
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Ali Aslaner, Attending Emergency Physician, Nevsehir Public Hospital
Other Study IDs: NevsehirPH
Record Dates: First submitted 2016-12-25; First posted 2017-02-02 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Altered Level of Consciousness
Keywords: documentation; altered mental status; definition; clinically
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Altered mental status (AMS) is common in older patients. However there is a lack of standardization in the definition and documentation of this compliant. Different perception of AMS can cause negative impact on interpretation and obtaining scientific data. Although definition of AMS is so complicated, clinical documentation can be detected in these patients with AMS.

DETAILED DESCRIPTION:
Basically, consciousness is the state of full awareness of the self and one's relationship to the environment. There are 2 related areas of neurologic function that are connected to consciousness: content (orientation and memory) and level (arousal and response to stimuli).

The mental changes are best looked for in terms of arousal, attention, alertness, orientation, cognition, memory, affect, and perception. Arousal (level of consciousness) can be detected by the Richmond Agitation and Sedation Scale. Others are related to content of consciousness and can be evaluated by cognitive tests. After one month pilot study, the investigators chose 5 features of content of consciousness due to easy applicable and detectable;

1. Attention (counting numbers backwards from 20) (>1 error positive)
2. Cognition (disorganized thinking; meaningless speech, irrelevant explanations)
3. Perception (visual or auditory hallucinations)
4. Memory (3 items recall) (>1 error positive)
5. Orientation (day of week, month and year) (>1 error positive)

These features are also combination of six item screener test and delirium symptoms.

All elderly patients (65 aged and older) presented to the emergency department, will be assessed according to these two methods; content and level of consciousness. And also, every patient's baseline status of consciousness will be obtained from surrogates who knows the patient best. All changes from patient's baseline status will be recorded. The investigators will investigate how changes are reflected in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* All older ED patients

Exclusion Criteria:

* Unknown baseline status, any trauma, and unable to assess mental status due to acute clinical condition (STE MI, severe dyspnea, etc)

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All older emergency department patients aged 65 and older.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06

PRIMARY OUTCOMES:
Detection of impaired level of consciousness in older ED patients | First 30 minute of presentation to the emergency department
  Arousal (level of consciousness) measured by the Richmond Agitation and Sedation Scale.
Detection of impaired content of consciousness in older ED patients | First 30 minute of presentation to the emergency department
  Awareness (content of consciousness) measured by the 5 criteria list questionnaire.

SECONDARY OUTCOMES:
Mortality | 1 and 3 month mortality after patient enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Nevsehir State Hospital, Nevşehir, Turkey (Türkiye)

REFERENCES:
- [Background] Aslaner MA, Boz M, Celik A, Ahmedali A, Eroglu S, Metin Aksu N, Eroglu SE. Etiologies and delirium rates of elderly ED patients with acutely altered mental status: a multicenter prospective study. Am J Emerg Med. 2017 Jan;35(1):71-76. doi: 10.1016/j.ajem.2016.10.004. Epub 2016 Oct 5. PMID 27765479
- [Background] Han JH, Wilber ST. Altered mental status in older patients in the emergency department. Clin Geriatr Med. 2013 Feb;29(1):101-36. doi: 10.1016/j.cger.2012.09.005. PMID 23177603
- [Background] European Delirium Association; American Delirium Society. The DSM-5 criteria, level of arousal and delirium diagnosis: inclusiveness is safer. BMC Med. 2014 Oct 8;12:141. doi: 10.1186/s12916-014-0141-2. PMID 25300023